CLINICAL TRIAL: NCT06984497
Title: Efficacy and Safety of Different Transplantation Routes of Human Umbilical Cord-mesenchymal Stem Cells in Patients With End-stage Liver Disease
Brief Title: Human Umbilical Cord-mesenchymal Stem Cells Via Different Transplantation Routes in ESLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHNKKY-DRSC
Record Dates: First submitted 2025-05-12; First posted 2025-05-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: End-Stage Liver Diseases
Keywords: cirrhosis; end-stage liver diseases; umbilical cord-mesenchymal stem cells; randomized controlled trial
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peripheral veins infusion group (Experimental): Peripheral veins infusion of stem cells
  Interventions: Other: Infusion of umbilical cord-mesenchymal stem cells through peripheral veins
- Hepatic arterial infusion group (Experimental): Hepatic arterial infusion of stem cells
  Interventions: Other: Infusion of umbilical cord-mesenchymal stem cells through hepatic artery

INTERVENTIONS:
Other: Infusion of umbilical cord-mesenchymal stem cells through peripheral veins — Umbilical cord-mesenchymal stem cells injected through peripheral veins
  Arms: Peripheral veins infusion group
Other: Infusion of umbilical cord-mesenchymal stem cells through hepatic artery — Umbilical cord-mesenchymal stem cells injected through hepatic artery
  Arms: Hepatic arterial infusion group

SUMMARY:
Stem cells are non-terminal cells that can self renew and replicate through symmetric or asymmetric division, with the potential to differentiate into different types of cells and tissues. Multiple studies have shown that human umbilical cord mesenchymal stem cell has good safety and effectiveness in improving acute or chronic liver injury.

Stem cell therapy for end-stage liver disease (ESLD) can be administered through various routes, among which hepatic artery and peripheral vein infusions are the most commonly used in clinical practice. The efficacy of hepatic artery infusion appears to be greater than that of peripheral vein infusion.

DETAILED DESCRIPTION:
Thirty-two participants with end-stage liver disease admitted to the Department of Gastroenterology of the General Hospital of Northern Theater Command are expected to be enrolled over a period of 6 months. They will be randomly assigned to peripheral vein infusion and hepatic arterial infusion of human umbilical cord mesenchymal stem cell groups. The investigators will observe alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, albumin, prothrombin time, international normalized ratio, model for end-stage liver disease score, and Child-Pugh score at weeks 4, 12, and 24 post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old

   -
2. End-stage liver disease

   -
3. Signed informed consent

Exclusion Criteria:

1. Tumours of the liver or other organs

   -
2. Liver transplantation recipients

   -
3. Acute myocardial infarction, acute heart failure, type I and type II respiratory failure, pulmonary embolism, acute cerebral infarction, acute cerebral haemorrhage and other serious cardiopulmonary diseases

   -
4. Other diseases that may seriously affect the survival

   -
5. Human immunodeficiency syndrome

   -
6. Interferon or glucocorticoid therapy within 1 year

   -
7. Treated for mental illness

   -
8. Participation in other clinical trials within 30 days

   -
9. Pregnant or breastfeeding subjects

   -
10. Allergic asthma, allergic urticaria, eczema, or a history of multiple drug and food allergies

    -
11. Other circumstances that are unsuitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 24 weeks
  Number of subjects surviving after 24 weeks

SECONDARY OUTCOMES:
Changes in Model for End-Stage Liver Disease (MELD) score | 4, 12, and 24 weeks
  The Model for End-Stage Liver Disease (MELD) score ranges from 6 to 40, with higher values indicating more severe liver dysfunction and an increased risk of mortality.
Changes in Child-Pugh score | 4, 12, and 24 weeks
  The Child-Pugh score is categorized into class A (5-6 points), class B (7-9 points), and class C (≥10 points), reflecting progressive liver disease severity. Higher Child-Pugh scores are associated not only with increased mortality risk but also with a significantly higher incidence of complications, such as gastrointestinal bleeding and infections.
Incidence of hepatic decompensation events | 4, 12, and 24 weeks
  Number of patients who developed gastrointestinal bleeding, ascites, and hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, MD, Study Director — The General Hospital of Northern Theater Command Study Director; Beilei Zhang, MM, Principal Investigator — The General Hospital of Northern Theater Command Study Director
Locations (1):
- General Hospital of Northern Theater Command Recruiting, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyra AC, Soares MB, da Silva LF, Braga EL, Oliveira SA, Fortes MF, Silva AG, Brustolim D, Genser B, Dos Santos RR, Lyra LG. Infusion of autologous bone marrow mononuclear cells through hepatic artery results in a short-term improvement of liver function in patients with chronic liver disease: a pilot randomized controlled study. Eur J Gastroenterol Hepatol. 2010 Jan;22(1):33-42. doi: 10.1097/MEG.0b013e32832eb69a. PMID 19654548
- [Background] Zhou GP, Jiang YZ, Sun LY, Zhu ZJ. Therapeutic effect and safety of stem cell therapy for chronic liver disease: a systematic review and meta-analysis of randomized controlled trials. Stem Cell Res Ther. 2020 Sep 25;11(1):419. doi: 10.1186/s13287-020-01935-w. PMID 32977828